CLINICAL TRIAL: NCT04632160
Title: A Study to Evaluate the Corvia Medical, Inc. IASD® System II to REDUCE Elevated Left Atrial Pressure in Patients With Heart Failure
Brief Title: Extended IASD Investigation: REDUCE LAP-HF IV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn pending formal analysis of REDUCE LAP-HF II Pivotal Study results
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001
Record Dates: First submitted 2020-11-06; First posted 2020-11-17 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment arm will undergo a fluoroscopically and intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) guided trans-septal puncture and IASD System II implant procedure.
  Interventions: Device: IASD System II

INTERVENTIONS:
Device: IASD System II — The implant is placed across the interatrial septum using a percutaneous transcatheter approach.
  Other Names: Interatrial Shunt Device

SUMMARY:
Multicenter, Prospective, Open Label, Single Arm, Clinical Trial.

The primary objective of this clinical trial is to further evaluate the safety and clinical efficacy of the IASD System II in symptomatic heart failure patients with an left ventricular ejection fraction (LVEF) ≥ 40%, and elevated left sided filling pressures despite standard Guideline Directed Medical Therapy (GDMT); and to compare the safety and efficacy results to those from the treatment arm of the REDUCE LAP-HF Randomized Trial II (Corvia protocol 1601).

DETAILED DESCRIPTION:
Participants are screened against non-invasive eligibility criteria and scheduled for a hemodynamic evaluation. Following right heart catheterization at rest and during supine bicycle exercise, patients will undergo a brief intracardiac echocardiography (ICE) or transesophageal echocardiography (TEE) exam for septal suitability.

Eligible patients continue with, fluoroscopically and echo guided transseptal puncture and IASD System II implant procedure. If a previously unknown protocol exclusion is discovered during the index procedure, and device is not implanted, participant is followed for 30 days, and then exits the study.

Participants return for follow-up exams 30 days after the implant procedure and annually for 5 years after the implant procedure. In-person visits will take place for the first 2 years. Telephone follow-up and medical chart review will be conducted for years 3-5.

ELIGIBILITY:
Select Inclusion Criteria:

* Chronic symptomatic heart failure with preserved or mid-range left ventricular ejection fraction (HFpEF or HFrEF)
* Participant is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams

Select Exclusion Criteria:

* Myocardial infarction and/or percutaneous cardiac intervention within past 3 months; Coronary artery bypass surgery in past 3 months, or current indication for coronary revascularization; AVR (surgical AVR or TAVR) within the past 12 months
* Advanced heart failure
* History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within the past 6 months
* Significant heart valve disease
* Chronic pulmonary disease
* Women of childbearing potential
* Severe obstructive sleep apnea not treated with CPAP or other measures

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of and time-to-cardiovascular mortality or first non-fatal, ischemic stroke through 12 months | 12 Month
Total rate (first plus recurrent) per patient year of heart failure (HF) admissions or healthcare facility visits for IV diuresis for HF up to 24 months, analyzed when the last subject completes 12 month follow-up, and time-to-first HF event | Up to 24 Months
Change in baseline Kansas City Cardiomyopathy Questionnaire (KCCQ) total summary score at 12 months | 12 Month

SECONDARY OUTCOMES:
Cardiovascular mortality through 12 months | 12 Months
Non-fatal, ischemic stroke through 12 months | 12 Months
New onset or worsening of kidney dysfunction (defined as eGFR decrease of > 20 ml/min/1.73 m2) through 12 months | 12 Months
Incidence of Major Cardiac Events i. Cardiac death ii. Myocardial infarction iii. Cardiac tamponade iv. Emergency cardiac surgery. | 12 Months
Thrombo-embolic complications (TIA, systemic embolization) through 12 months | 12 Months
≥30% increase in right ventricular size/decrease in TAPSE through 12 months | 12 Months
Newly acquired persistent or permanent AF or atrial flutter through 12 months | 12 Months
Total rate per patient year of heart failure admissions or healthcare facility visits for IV diuresis or visits with intensification of oral diuresis for HF through 24 months, analyzed when the last subject completes 12 months follow-up | Up to 24 months
Change in New York Heart Association (NYHA) functional Class between baseline and 12 months | 12 Months
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score between baseline and 12 months, categorized as ≤0, >0 - 5, >5 - 10, >10 - 15, >15 - 20, >20 - 25, >25. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sanijv Shah, MD, Principal Investigator — Northwestern Memorial Hospital; Marty Leon, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No